

# Non-Interventional Study Protocol <B0661178>

# Safety and effectiveness of apixaban compared to warfarin in NVAF patients at higher risk of bleeding

Statistical Analysis Plan (SAP)

Version: Ver.1

Author: PPD

**Date**: 29-Jun-2022

# **TABLE OF CONTENTS**

| 1. | AMENDMENTS FROM PREVIOUS VERSION(S) | 4 |
|---|---|---|
| 2. | INTRODUCTION | 4 |
| 3. | STUDY DESIGN | 5 |
| 3.<br>3.<br>3. | Data source | 6 |
| 3. | | |
| | .4.1. The research questions: | |
| 4. | HYPOTHESES AND DECISION RULES | |
| 4.<br>4.<br>4.<br>4. | STATISTICAL HYPOTHESES STATISTICAL DECISION RULES ANALYSIS SETS/POPULATIONS FULL ANALYSIS SET .4.1. Inclusion criteria .4.2. Exclusion criteria | |
| 5. | .4.3. Definitions | |
| <b>6.</b> | OTHER ANALYSIS SET | |
| 7. | SUBGROUPS | |
| 8. | ENDPOINTS AND COVARIATES | |
| 8.<br>8. | EFFICACY/EFFECTIVENESS ENDPOINT(S) | 11 |
| 9. | OTHER ENDPOINTS | 13 |
| 10. | COVARIATES | 13 |
| 11. | HANDLING OF MISSING VALUES | 16 |
| 12. | STATISTICAL METHODOLOGY AND STATISTICAL ANALY | SES 16 |
| 12 | 2.1.1. Calculation of Propensity Score 2.1.2. Inverse probability treatment weighting (IPTW) | 16<br>17<br>18<br>not defined. |
| | 2.1.5. Exploratory subgroup analysis | 19 |

| | 12.1.6.<br>12.1.7.<br>12.1.8.<br>12.1.9.<br>12.1.10. | Analysis of Continuous Data | ned<br>. 19<br>. 19 |
|---|---|---|---|
| 13. | LIST | OF TABLES AND TABLE SHELLS | . 20 |
| 14. | REFE | CRENCES | . 20 |
| 15. | APPE | NDICES | . 27 |
| 1 | 5.2. AP | PENDIX 1: DATA DERIVATION DETAILSPENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS . PENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY | 27 |
| 16. | EFFE | CTIVENESS ENDPOINTS | . 43 |
| <b>17.</b> | SAFE | TY ENDOPOINTS | . 44 |
| 18. | BLEE | CDING | . 45 |
| 10 | VARI | ARI ES FOR SURCROUP ANALYSIS | <b>5</b> 1 |

# 1. AMENDMENTS FROM PREVIOUS VERSION(S)

Not applicable since this is the first version and no amendment

#### 2. INTRODUCTION

Atrial fibrillation (AF) is characterized by a rapid, irregular heartbeat which can cause blood to pool in the atria and increase the risk of the formation of blood clots. AF affects 0.6% to 1.6% of the general population and up to 14% in cardiovascular clinics in Japan<sup>1-3</sup>. AF can be categorized into three main categories based on patient characteristics: lone atrial fibrillation – AF in the absence of overt cardiovascular disease or precipitating illness non-valvular AF (NVAF) – presence of AF without concurrent rheumatic mitral valve disease or history of mitral valve repair or prosthetic heart valve; and secondary AF-AF that occurs in the setting of acute myocardial infarction (MI), cardiac surgery, pericarditis, myocarditis, hyperthyroidism, pulmonary embolism, pneumonia, or other acute pulmonary disease. Anticoagulation therapy is important to prevent thromboembolism in patients with NVAF. Warfarin, a vitamin K antagonist, is the first oral anticoagulant approved for the treatment and prevention of thromboembolism in Japan in 1962 and it had long been the only oral anticoagulant until the first non-vitamin K antagonist oral anticoagulants (NOACs), dabigatran, was introduced with approval for NVAF treatment in March  $2011^4$ . Apixaban was approved in December 2012 in Japan and demonstrated superiority compared to warfarin in preventing stroke or systemic embolism, caused less bleeding, and resulted in lower mortality in patients with atrial fibrillation in Phase 3 clinical trial<sup>5</sup>.

Although randomized control trials (RCTs) aimed at head-to-head comparison with placebo or a reference drug may provide evidence of safety and efficacy of treatments at the highest level, there are potential limitations derived from a limited number of pre-selected patients and strict patient eligibility criteria with regard to age, comorbidities, and concomitant medications. Accordingly, these studies may not accurately represent what happens when drugs are used in general clinical practice. Especially data for Japanese NVAF patients are limited due to limited number of Japanese patients recruited in the RCT. Also patients with higher risk from a safety perspective, for instance patients with active caner, are generally excluded from RCT and further limited data are existed. Previously we have shown that bleeding risks as well as stroke/SE risks are less in real world clinical practice in Japan compared to warfarin<sup>6-8</sup>, but there are still little data for Japanese NVAF patients who has higher bleeding risks such as components of HAS-BLED risk score factors, active cancer, uncontrolled hypertension etc. The objectives of this study is to compare the risk of incidence of

stroke and bleeding among NVAF patients with such higher bleeding risk(s) newly prescribed

apixaban or warfarin using a nation-wide administrative claims database.

#### 2.1. STUDY DESIGN

This is a retrospective observational study using data from Medical Data Vision Co. Ltd. (MDV Co. Ltd.) database (data set from 1 March, 2011 to 31 Jun, 2021). Among patients registered in the database, patients are selected based on the inclusion and exclusion criteria (see below).

Study measures include: (1) for safety evaluation: major bleeding (primary safety endpoint, defined as any bleeding requiring hospitalization for treatment); (2) for effectiveness evaluation: a composite of ischemic stroke, hemorrhagic stroke or SE (primary effectiveness endpoint).

The primary purpose of this study is to investigate the safety and effectiveness of apixaban compared to warfarin in patients who are prone to bleeding, with at least one known risk factor for bleeding. The analyses will be conducted using the 3-step procedure shown below,

First, all patients with NVAF who are newly diagnosed and initiated apixaban or warfarin will be extracted from the database. Among these patients, patients with at least one predetermined high bleeding risks will be extracted. In this study, predetermined high bleeding risks are 1) patients with hypertension diagnosis, 2) patients with liver dysfunction, 3) patients with renal dysfunction diagnosis, 4) patients with a history of bleeding, 5) patients with hemorrhagic stroke, 6) patients with alcohol abuse, 7) patients with concomitant used of antiplatelet drugs, 8) patients with chronic (continuously for longer than 90 days) concomitant use of Non-steroidal antiinflammatory drug (NSAID), 9) highly elderly (> 80 years old), 10) patients with refractory hypertension, 11) patients with a history of peptic ulcer diagnosis, 12) patients with active cancer, 13) patients with diabetes mellitus, 14) patients whose body weight is <40kg, 15) patients with polypharmacy (sea Section 5.4 for the definition). Patients with at least one predetermined high bleeding risk factor will be divided into two cohorts, apixaban and warfarin cohorts, based on the first prescribed drug just after the NVAF diagnosis. Patient characteristics will be balanced by using an inverse probability of treatment weighting (IPTW) method to create balanced apixaban and balanced warfarin cohorts. Comparisons will be conducted by using these balanced warfarin and apixaban cohorts (Kaplan-meier curves, incidence rates per 1,000 person-year and hazard ratio with 95% confident intervals). The primary safety and effectiveness analyses are comparison of apixaban with warfarin in patients with at least one predetermined risk factor for bleeding.

- Second, after the first analysis, we will conduct separate interaction analysis of the treatment (apixaban vs. warfarin) and one of the 15 risk factors (e.g., hypertension yes vs no, etc) to see if treatment effects are consistent among patients with or without each specific factor
- Third, patients will be stratified by risk factors into 15 subgroups, and same IPTW analyses as described in the step 1 will be conducted only in the subgroups with adequate sample sizes.

The follow-up period is variable, and will begin on the next day of the index date and continue until the earliest of the following scenarios – occurrence of target outcome event (details available in Subsection 5); discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database.

### 2.1.1. Study population

The study population will consist of adults with NVAF who are newly prescribed apixaban or warfarin with at least one high bleeding risk. Further information on patient selection and enrolment and follow-up time periods are available in Subsection 9.2 of the protocol.

#### 2.1.2. Data source

The analysis will be based on administrative data from MDV Co. Ltd., a longitudinal database based on health insurance claims and medical records obtained from the hospitals in which the DPC payment system for utilization of both inpatient and outpatient hospital claims (percentage of inpatients is about 20%). The database provides claims data from 449 hospitals (as of Aug 2021) using the DPC system for medical service claims (26% of general hospitals in Japan is under the DPC system) including approximately 36.7 million patient data.

#### 2.1.3. Treatment/cohort labels

For primary analysis,

- IPTW-balanced apixaban cohort: NVAF patients de novo diagnosis with NVAF and initiate apixaban and have at least one risk factor(s) of bleeding.
- IPTW-balanced warfarin cohort: NVAF patients de novo diagnosis with NVAF and initiate warfarin and have at least one risk factor(s) of bleeding.

Patients will be assigned to each cohort based on the first prescription of oral anticoagulants after the diagnosis of NVAF (warfarin or apixaban). If the 1<sup>st</sup> prescribed oral anticoagulants are not warfarin

nor apixaban, the patients will be excluded. Patient clinical and demographic characteristics will be balanced by using IPTW methods.

#### 2.2. STUDY OBJECTIVES

#### 2.2.1. The research questions:

- 1. Are there any differences in the risk of major bleeding between apixaban and warfarin for patients with higher bleeding risk(s) in the general practice settings in Japan?
- 2. Are there any differences in the risk of stroke/systemic embolism(SE) between apixaban and warfarin for patients with higher bleeding risk(s) in the general practice settings in Japan?

### 2.2.2. The primary objective of the study

To compare effectiveness (a composite risk of stroke/SE) and safety (major bleeding events) of warfarin and apixaban among NVAF patients with at least one bleeding risk (that is, patients at higher risk of bleeding)

#### 2.2.3. The secondary objectives are

- 1. To compare the risk of major gastrointestinal or intracranial bleeding between warfarininitiators and apixaban-initiators in patients with at least one bleeding risk.
- 2. To compare the risk of ischemic stroke, hemorrhagic stroke or SE between warfarin-initiators and apixaban-initiators in patients with at least one bleeding risk.

F

#### 2.2.4. Objectives of other exploratory analysis are

To explore the risk of major bleeding and stroke/SE in the specific populations at higher bleeding risk(s).

As shown above (see 2.1), after interaction analyses of the treatment and risk factors, patients will be stratified to subgroups by each of above mentioned 15 predetermined risk factors separately. Subgroups with adequate sample size will be selected for IPTW analyses.

In the previous feasibility analysis, we found that the numbers of patients with hemorrhagic stroke, alcohol abuse, chronic concomitant used of NSAIDs (for continuously > 90 days), and refractory hypertension were less than 2,000. Due to the insufficient statistical power, these subgroups could be eliminated from the further subgroup analysis. Again, the final decision will be based on the formal evaluation of the number of sample sizes N in those subgroups.

Candidates of exploratory subgroups listed based on the preliminary feasibility analysis

- - Exploratory analysis regarding hypertension
  - Exploratory analysis regarding liver dysfunction.
  - Exploratory analysis regarding renal impairment.
  - Exploratory analysis regarding bleeding including intracranial hemorrhage
  - Exploratory analysis regarding concomitant use of antiplatelet drug
  - Exploratory analysis by age
    - $\checkmark$  > 80 y
    - $\checkmark$  > 90 y
  - Exploratory analysis regarding peptic ulcer
  - Exploratory analysis regarding active cancer
  - Exploratory analysis regarding low body weight (<40kg)
  - Exploratory analysis regarding diabetes mellitus
  - Exploratory analysis regarding polypharmacy (≥6 medicines)

#### 3. HYPOTHESES AND DECISION RULES

#### 3.1. STATISTICAL HYPOTHESES

This study includes specific hypotheses to be tested. The null hypothesis for each objective is as follows:

Null: The risks of each of the following endpoints do not differ between NVAF patients treated with warfarin and patients treated with apixaban even if the patients have at least one bleeding risk.

- Major Bleeding
- A composite of stroke/SE

#### 3.2. STATISTICAL DECISION RULES

For primary safety and effectiveness analyses, all statistical tests will be performed at p=0.05 (two-sided) with no adjustment for multiplicity. Since we will conduct various multiple subgroup analyses, which lead to the "Multiple Testing Problem". Here these subgroup analyses will be conducted with an exploratory purpose and we do not plan to conclude anything from the results here. Therefore, we will not adjust the p values and still the use p<0.05 to indicate the statistical significance.

#### 4. ANALYSIS SETS/POPULATIONS

#### 4.1. FULL ANALYSIS SET

This study uses data from the MDV database, which includes the data used for both inpatient and outpatient insurance claims by hospitals according to the Diagnosis Procedure Combination (DPC) procedure.

The study population will consist of adults with NVAF who are newly prescribed apixaban or warfarin. Follow-up time period starts from the next day of the index date, and ends depending on following outcomes which observed first.

#### 4.1.1. Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Patients with diagnosis with NVAF anytime in the baseline period or on the index date,
- 2. The first prescribed anticoagulant is apixaban or warfarin after the index date.
- 3. No use of the any oral anticoagulants (OACs) during the baseline period (the 180 days before the index date)
- 4. Age of 18 years or older on the index date.

#### 4.1.2. Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

- 1. Having a diagnosis of valvular atrial fibrillation, post-operative atrial fibrillation, rheumatic atrial fibrillation or mechanical-valvular atrial fibrillation during the baseline and post-index period
- 2. Having a procedure of prosthetic heart valve during the baseline period
- 3. Having a cardiac surgery procedure record during the baseline period
- 4. Having a diagnosis of venous thromboembolism during the baseline period
- 5. Having a hemodialysis during the baseline period
- 6. Female patients with pregnancy during the baseline and follow-up period
- 7. Patients prescribed apixaban other than approved daily dose (<5 mg or >10 mg)
- 8. Patients prescribed OACs during baseline period

#### 4.1.3. Definitions

#### 4.1.3.1. Follow-up period

Follow-up time period starts from the next day of the index date, and ends depending on following outcomes which observed first.

- 1. Major bleeding when the target outcome for the analysis is major bleeding.
- 2. Composite of (ischemic or hemorrhagic) stroke and SE when the target outcome for the analysis is the composite endpoint.
- 3. Discontinuation of apixaban or warfarin: The index treatment will be considered to be "discontinued" if apixaban or warfarin is not prescribed within 45 days after prescription refill date (calculated from the last refill date plus days of supply) of apixaban or warfarin, even though the patient has >1 medical encounter records after more than 45 days following the prescription refill date. The supposed prescription refill date is regarded as the last day of the follow-up for discontinued patients.
- 4. Switching from apixaban or warfarin: The index treatment is regarded as "switched" if the OAC is prescribed within 45 days after prescription refill date of apixaban or warfarin when the patient has 1> medical encounter records after more than 45 days following the prescription refill date. The switched day is regarded as the last day of the follow-up for the switched patients.
- 5. Withdrawal from the database: The patients are regarded as "withdrawal" from the database if apixaban or warfarin is not prescribed within 45 days after prescription refill date of the apixaban or warfarin and there is no data of the patient on the database after prescription refill date. The last medical encounter is regard as the last day of the follow-up for patients withdrawn from the database.
- 6. An elapse of 2 years from the index date without any of the event above.

#### 4.1.3.2. Index date

The date when patients initiated warfarin or apixaban

#### 4.2. SAFETY ANALYSIS SET

Safety-related events other than bleeding will not be collected for this analysis. As mentioned above, bleeding will be investigated as safety-related primary endpoints. However, other adverse events,

•

serious AE or non-serious AE will not be collected in this analysis because the dataset provided by MDV will not contain the AE-related information.

#### 4.3. OTHER ANALYSIS SET

None

#### 4.4. SUBGROUPS

Following subgroups will be created and exploratory analyses for primary endpoints (major bleeding or stroke/SE) will be performed.

| Variable | categories |
|------------------------------------------------------|----------------------|
| Hypertension diagnosis | Yes or No |
| Liver dysfunction diagnosis | Yes or No |
| Renal impairment diagnosis | Yes or No |
| Bleeding diagnosis including intracranial hemorrhage | Yes or No |
| Treated with antiplatelet drug (>28d) | Yes or No |
| Ago | >80 years |
| Age | >90years |
| Peptic ulcer diagnosis | Yes or No |
| Cancer diagnosis | Yes or No |
| Low body weight | <40 kg |
| Diabetes mellitus diagnosis | Yes or No |
| Polypharmacy | ≥6 concomitant drugs |

#### 5. ENDPOINTS AND COVARIATES

# 5.1. EFFICACY/EFFECTIVENESS ENDPOINT(S)

| Variable | Role | Operational definition |
|---|---|---|
| Stroke/SE<br>(composite)<br>event after<br>index date | Outcome<br>(primary<br>endpoint) | Operational definition of Stroke and SE will follow the operational definition of Stroke event after index date and SE event after index date. Time to events will be defined as the number of days from the index date to the occurrence of the first stroke or SE. |
| Ischemic<br>stroke event<br>after index<br>date | Outcome<br>(secondary<br>endpoint) | Ischemic stroke after index date not including the index date will be identified using hospital claims which had an ischemic stroke diagnosis code as the first listed ICD-10 diagnosis code (Appendix, 10.3.3). An event occurrence of ischemic stroke is defined as a case that "01: Disease name which input the most medical resources", "02:Sub-disease name", "11: Main disease name", "21: Disease name behind hospitalization", or "31: Disease name which input the second most medical resources" in DPC database. Time to ischemic |

| Variable | Role | Operational definition |
|---|---|---|
| | | stroke will be defined as the number of days from the index date to the occurrence of the first ischemic stroke. |
| Hemorrhagic stroke event after index date Outcome (secondary endpoint) | | Hemorrhagic stroke after index date not including the index date will be identified using hospital claims which had a hemorrhagic stroke diagnosis code as the first listed ICD-10 diagnosis code (Appendix, 10.3.3). An event occurrence of hemorrhagic stroke is defined as a case that "01: Disease name which input the most medical resources", "02:Sub-disease name", "11: Main disease name", "21: Disease name behind hospitalization", or "31: Disease name which input the second most medical resources" in DPC database. Time to hemorrhagic stroke will be defined as the number of days from the index date to the occurrence of the first hemorrhagic stroke. |
| SE event after index date | Outcome<br>(secondary<br>endpoint) | SE after index date not including the index date will be identified using hospital claims which had a SE diagnosis code as the first listed ICD-10 diagnosis code (Appendix, 10.3.3). An event occurrence of SE is defined as a case that "01: Disease name which input the most medical resources", "02:Sub-disease name", "11: Main disease name", "21: Disease name behind hospitalization", or "31: Disease name which input the second most medical resources" in DPC database. Time to SE will be defined as the number of days from the index date to the occurrence of the first SE event. |

# 5.2. SAFETY ENDPOINTS

| Variable | Role | Operational definition |
|---|---|---|
| Major bleeding event after index date | Outcome<br>(primary<br>endpoint) | Major bleeding after index date will be identified using hospital claims which had a bleeding diagnosis code as the first listed ICD-10 or disease code (Appendix 10.3.5). An event occurrence of major bleeding is defined as a case that "21: Disease name behind hospitalization" in DPC database. Time-to-major bleeding will be defined as the number of days from the index date to the occurrence of the first major bleeding event. |
| Major ICH bleeding event after index date Outcome (secondary endpoint) | | Major ICH bleeding after index date will be identified using hospital claims which had an ICH bleeding diagnosis code as the first listed ICD-10 or disease code (Appendix, 10.3.4). An event occurrence of major bleeding is defined as a case that "21: Disease name behind hospitalization" in DPC database. Time-to-major ICH bleeding will be defined as the number of days from the index date to the occurrence of the first major ICH bleeding event. |
| Major GI<br>bleeding event<br>after index<br>date | Outcome<br>(secondary<br>endpoint) | Any GI bleeding after index date will be identified using hospital claims which had a GI bleeding diagnosis code as the first listed ICD-10 or disease code (Appendix, 10.3.4). Time-to-any GI bleeding will be defined as the number of days from the index date to the occurrence of the first any GI bleeding event. |

#### **5.3. OTHER ENDPOINTS**

None

# **5.4. COVARIATES**

Demographic and clinical characteristics are collected during the baseline period, at the index date or during follow-up period.

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Sex Category | Baseline characteristic | Index date | Dichotomous variable equals 1 if sex is male and 2 if female |
| Age | Baseline characteristic | Index date | Age (in years) at the index date |
| Age (> 80y, >90y) | Sub-group identifier | Index date | Age (in years) at the index date |
| Body weight | Baseline characteristic | Baseline<br>period | ≥ 60 kg or < 60 kg |
| eGFR (continuous) | Baseline characteristic | Baseline<br>period | Value in the baseline If a patient has multiple eGFR values, the values closest to the index date will be adopted If a patient does not have eGFR values, but has serum creatinine values, an eGFR value is |

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| | | | calculated from a serum creatinine value using fomulas. |
| eGFR (categorical) | Baseline characteristic | Baseline<br>period | ≥ 50 ml/min or < 50 ml/min<br>If a patient does not have eGFR values, but has<br>serum creatinine values, an eGFR value is<br>calculated from a serum creatinine value using<br>fomulas. |
| Serum creatinine<br>(continuous) | Baseline characteristic | Baseline<br>period | Value in the baseline If a patient has multiple eGFR values, the values closest to the index date will be adopted If a patient does not have serum creatinine values but has eGFR values, a serum creatinine value is calculated from eGFR value using fomulas |
| Serum creatinine<br>(categorical) | Baseline characteristic | Baseline<br>period | ≥ 1.5mg/mL or < 1.5 mg/mL If a patient does not have serum creatinine values but has eGFR values, a serum creatinine value is calculated from eGFR value using fomulas |
| CHADS2 | Baseline characteristic | Baseline<br>period | CHADS2 score will be calculated based on age and<br>the presence of congestive heart failure,<br>hypertension, diabetes, and stroke or TIA. |
| CHA2DS2-VASc | Baseline characteristic | Baseline<br>period | Score calculated by appointing 1 point each for congestive heart failure/left ventricle dysfunction, hypertension, diabetes, vascular disease (prior MI, peripheral arterial disease, or aortic plaque), age between 65-74, female gender; and 2 points each for age >75 years and prior stroke, TIA, or thromboembolism. |
| Heart failure<br>diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for heart failure ICD-10 or disease codes during the baseline period. |
| Coronary heart<br>disease diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for coronary heart disease ICD-10 or disease codes during the baseline period. |
| Peripheral arterial<br>disorder diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for peripheral arterial disorder ICD-10 or disease codes during the baseline period. |
| Myocardial infarction diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for myocardial infarction ICD-10 or disease codes during the baseline period. |
| Hyperthyroidism or thyrotoxicosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for hyperthyroidism ICD-10 or disease codes during the baseline period. |
| Stroke, TIA or SE<br>diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for Stroke, TIA or systemic embolism ICD-10 or disease codes during the baseline period. |
| Renal dysfunction<br>diagnosis | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for renal dysfunction ICD-10 or disease codes during the baseline period. |
| Liver dysfunction diagnosis | Baseline characteristic<br>Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for liver dysfunction ICD-10 or disease codes during the baseline period. |
| Bleeding diagnosis | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for bleeding ICD-10 or disease codes during the baseline period. |

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Hypertension<br>diagnosis | Baseline characteristic<br>Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for hypertension ICD-10 or disease codes during the baseline period. |
| Refractory<br>hypertension<br>diagnosis | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are prescriptions of ATC codes or receipt codes for all of the following 4 drugs during the baseline period; calcium channel blocker, ACE inhibitor/ARB, thiazide diuretics and MR antagonist/a-blocker/b-blocker |
| Diabetes mellitus<br>diagnosis | Baseline characteristic<br>Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for diabetes mellitus ICD-10 or disease codes during the baseline period. |
| Cancer diagnosis | Baseline characteristic<br>Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for diabetes mellitus ICD-10 or disease codes during the baseline period. |
| Treated with antiplatelet drug | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of antiplatelet drug ATC or receipt codes during the baseline period. |
| Treated with antiplatelet drug (>28 d) | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of antiplatelet drug ATC or receipt codes during the baseline period. |
| Treated with NSAIDs | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of NSAIDs ATC or receipt codes during the baseline period. |
| Treated with NSAIDs (>90 d) | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of NSAIDs ATC or receipt codes during the baseline period. |
| Treated with gastric secretion inhibitor | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of gastric secretion inhibitor drug ATC or receipt codes during the baseline period. |
| Treated with statin-<br>based drug | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of statin-based drug ATC or receipt codes during the baseline period. |
| Treated with anti-<br>hypertensives | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of anti-hypertensive ATC or receipt codes during the baseline period. |
| Treated with anti-<br>arrhythmics | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of anti-arrythmics ATC or receipt codes during the baseline period. |
| Treated with beta-<br>blockers | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of beta-blockers ATC or receipt codes during the baseline period. |
| Treated with heparins | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 prescriptions of heparins ATC or receipt codes during the baseline period. |
| Cardioversion | Baseline characteristic | Baseline<br>period | Dichotomous variable equals 1 if there is ≥1 operation of cardioversion receipt codes during the baseline period. |
| Alcohol abuse | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for Alcohol abuse ICD-10 or disease codes during the baseline period. |
| Bleeding diagnosis | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for major or any bleeding ICD-10 or disease codes during the baseline period |

| Variable | Role | Data source(s) | Operational definition |
|---|---|---|---|
| Peptic ulcer<br>diagnosis | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for peptic ulcer ICD-10 or disease codes during the baseline period |
| Hemorrhagic<br>stroke diagnosis | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥1 diagnoses for hemorrhagic stroke ICD-10 or disease codes during the baseline period |
| Low body weight (<40 kg) | Sub-group identifier | Baseline<br>period | Body weight during baseline period |
| Polypharmacy | Sub-group identifier | Baseline<br>period | Dichotomous variable equals 1 if there are ≥6 prescriptions of oral drug ATC or receipt codes during the baseline period. |
| PT-INR<br>(Prothrombin time-<br>international<br>normalized ratio) | potential confounder | Baseline<br>period | Continuous variable. * Only available for patients treated with warfarin |
| Physician specialty | potential confounder | Index date | Dichotomous variable equals 1 if a physician specialty on the index date is categorized into a cardiac specialty and 0 if others. Following specialties will be categorized as the cardiac specialty: cardiology stroke, cardiovascular surgery, pediatric cardiology, neurosurgery, cardiovascular medicine, and neurology. If there are ≥1 specialties but including the cardiac specialty, the physician specialty will be regarded as the cardiac specialty. |
| Hospital size (<500 beds or not) | potential confounder | Index date | Dichotomous variable equals 1 if hospital size on the index date is <500 beds and 0 if ≥500 beds. |
| Hospitalization status on index date | potential confounder | Index date | Dichotomous variable equals 1 if hospitalization status is inpatient and 0 if outpatient. |
| INR (warfarin cohort) | Baseline characteristic | Baseline<br>period | Continuous variable. * Only available for patients treated with warfarin |
| Apixaban dose (2.5 g BID) | Baseline characteristic | Baseline<br>period | 2.5 mg BID or 5mg BID * Only available for patients treated with apixaban |

#### 6. HANDLING OF MISSING VALUES

Patients without all required data will be excluded from the analysis.

#### 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 7.1. STATISTICAL METHODS

#### 7.1.1. Calculation of Propensity Score

In this study, balanced cohorts (apixaban vs. warfarin) will be created by an IPTW method. Propensity scores will be estimated by unconditional logistic regression analyses that incorporate potential predictors of therapy as independent variables in the regression and cohort status as the outcome. Using calculated propensity score an IPTW method will be applied to balance the warfarin and apixaban cohorts, which will be used for the comparisons of all endpoints (sections 5.1 and 5.2). The following covariates will be included in the logistic regression for calculation of propensity score:

• age on index date

- gender
- CHADS2 score in baseline
- CHA2DS2-VASc score in baseline
- heart failure diagnosis in baseline
- coronary heart disease diagnosis in baseline
- peripheral arterial disorder diagnosis in baseline
- myocardial infarction diagnosis in baseline
- hyperthyroidism or thyrotoxicosis in baseline
- TIA diagnosis in baseline
- stroke or SE diagnosis in baseline
- renal dysfunction diagnosis in baseline
- liver dysfunction diagnosis in baseline
- bleeding diagnosis in baseline
- hypertension diagnosis in baseline
- diabetes mellitus diagnosis in baseline
- treated with antiplatelet drug in baseline
- treated with NSAIDs in baseline
- treated with gastric secretion inhibitor in baseline
- treated with statin-based drug in baseline
- treated with anti-hypertensives in baseline
- treated with anti-arrhythmics in baseline
- treated with beta-blockers in baseline
- treated with heparins in baseline
- cardioversion in baseline

The operational definitions for the above covariates are shown in the Section 5.4.

#### 7.1.2. Inverse probability treatment weighting (IPTW)

IPTW with stabilized weights will be used to balance patient characteristics between two groups using propensity score calculated by using a multivariable logistic model as mentioned above (see above 7.1.2.1). However, if a treated patient has a very low propensity score, a very large weight can be created, which leads to increased variability of the estimated treatment effect. In order to address this, the weights can be stabilized by using a formula shown below, by multiplying the treatment and control weights by a constant, equal to the expected value of being in the treatment or comparison cohorts, respectively.

 $W_i = \frac{Z}{PS_i} + \frac{1-Z}{1-PS_i}$ , z: probability of treatment without considering covariates

The distribution of the stabilized weight will be reviewed. If there are extreme outliers, the large weights could be set to a less extreme value (e.g. recoding all weights that are outside 5th and 95th percentile). If needed, truncation can be done after stabilizing the weights. After the weights are applied, the balance of the baseline covariates will be assessed. First, the means and proportions of baseline variables are compared. The standardized difference compares the difference in means in units of the standard deviation. If the standardized difference is less than 10%, the covariates are considered balanced.

#### 7.1.3. Analysis of Continuous Data

Continuous data will be summarized using descriptive statistics, including the mean, standard deviation, median, first and third quartiles, and minimum and maximum. Baseline characteristics (before and after IPTW weighting) will be compared between patients treated with warfarin and patients treated with apixaban, using the standardized difference.

#### 7.1.4. Analysis of Categorical Data

Counts and percentages will be provided for dichotomous and polychotomous variables of baseline patient characteristics when performing descriptive analysis. Standardized difference will be calculated for each variable (before and after IPTW weighting). For calculation of standardized differences, categorical variables will be converted into a set of binary indicators, one for each non-reference level of the variable.

#### 7.1.5. Kaplan-Meier Method

For each endpoint, Kaplan-Meier curves will be plotted for the time from the index date to first event by index OAC treatment in each of the propensity-score-weighted cohorts. The log-rank test will be used for comparison between two curves.

#### 7.1.6. Cox proportional hazards model

Cox proportional hazards model will be used to compare endpoints (time-to-endpoint) in the propensity-score-weighted cohorts with robust sandwich estimates to account for the potential clustering within weighted sets. The Cox proportional hazards model will include only index OAC treatment as the independent variable if patient characteristics are balanced between groups... If not balanced, the unbalanced variable will be also included to the model in addition to the index OAC PFIZER CONFIDENTIAL

treatment. The hazard ratios with corresponding 95% confidence intervals and p-values will be reported.

#### 7.1.7. Exploratory subgroup analysis

For subgroup analyses, hazard ratios with 95% confident intervals (95% CI) will be calculated using the Cox proportional hazards model as in primary analysis. As mentioned above, subgroup analyses are exploratory, no definitive conclusions from these subgroup analyses would be drawn.

#### 7.1.8. Sensitivity analysis

For the primary effectiveness and safety analysis, E-values<sup>10</sup> (evidence for causality) will be calculated based on calculated hazard ratios and 95% confident intervals to assess the extent of unmeasured confounding. The E-value is defined as the minimum strength of association for an unmeasured confounder with both the treatment and the outcome to explain away the observed significant (if any) treatment-outcome association.

#### 7.1.9. Power calculation

Incidence rates of stroke/SE and major bleeding in the primary analysis population here (that is, de novo NVAF patients initiating an anticoagulant therapy with warfarin or apixaban who have at least one bleeding risk factor) have not been investigated yet and hazard ratios of stroke/SE and major bleeding in apixaban users relative to warfarin users also have not been investigated yet. Therefore, we estimated the needed sample size to achieve adequate statistical power (e.g., 0.80) based on the major previous RCT and RWE conducted so far.

Stroke/SE

| Study | Subgroup | HR | Incidence rate<br>(%/year) | |
|---|---|---|---|---|
| | | | Warfarin | Apixaban |
| ARISTOTLE | - | 0.79 | 1.60 | 1.27 |
| | ≥ 75 years | | 2.2 1.6 | |
| | ≤ 60kg | | 3.2 2.0 | |
| | Prior stroke or TIA | | 3.2 2.5 | |
| | Diabetes | | 1.9 | 1.4 |
| | Severe to moderate renal dysfunction | | 2.7 | 2.1 |
| | Aspirin | | 1.9 1.3 | |
| CER3 | | 0.66 | 2.87 | 1.55 |

| ≥ 80 years | 4.04 | 2.06 |
|--------------------------------------|------|------|
| < 60 kg | 3.47 | 2.45 |
| Severe to moderate renal dysfunction | 2.50 | 1.33 |
| Anti-platelet | 3.61 | 1.93 |

Major bleeding

| Study | Subgroup | HR | | nce rate<br>year) |
|---|---|---|---|---|
| · | | | Warfarin | Apixaban |
| ARISTOTLE | - | 0.69 | 3.09 | 2.13 |
| | ≥ 75 years | | 5.2 | 3.3 |
| | ≤ 60kg | | 3.0 | 2.1 |
| | Prior stroke or TIA | | 3.9 | 2.8 |
| | Diabetes | | 3.1 | 3.0 |
| | Severe to moderate renal dysfunction | | 6.4 | 3.2 |
| | Aspirin | | 3.7 | 2.7 |
| CER3 | | 0.74 | 2.81 | 1.69 |
| | ≥ 80 years | | 3.94 | 2.35 |
| | < 60 kg | | 3.67 | 2.61 |
| | Severe to moderate renal dysfunction | | 3.32 | 2.21 |
| | Anti-platelets | | 3.07 | 1.91 |

As shown in Tables above, absolute incidence rates of stroke/SE and major bleeding could be higher in patients with (a) risk factor(s) associated with bleeding. However, the ARISTOTLE study has revealed that P-value for interaction was mostly >0.05 and relative risk (HR) may not be changed in the specific subgroups compared to the entire cohorts

Based on the incidence rates and HRs shown above, sample size required for adequate statistical power (e.g., power=0.8) was estimated as follows,

#### Sample size calculation

| Assumption:<br>Values used for<br>calculation | Calculated results |
|---|---|
| 0.05 | |
| 0.2 | |
| 0.7 | |
| 1:1 | |
| 3.77%/year** | |
| 2.50%/year** | |
| | 246*** |
| | 7,846 |
| | Values used for calculation 0.05 0.2 0.7 |

For Stroke/SE 0.05 Type I error rate Type II error rate 0.2 Hazard ratio\* 0.7 N ratio in apixaban and 1:1 warfarin cohorts 2.77%/year\*\* **Event rate for warfarin** Event rate for apixaban 1.79%/year\*\* **Total events needed** 246\*\*\* **Estimated number of patients** 10,789

In the preliminary check to examine the feasibility of this study, we have obtained that the number of apixaban users and of warfarin users who were eligible for this study were both more than 10,000 patients. Considering that IPTW will be applied to balance the patient characteristics in this study, the number of patients eligible for this study would be adequate for the primary analysis.

#### 7.2. STATISTICAL ANALYSIS

See sections  $2\sim5$ .

#### 7.2.1. Safety Analysis

See sections  $2\sim5$ .

#### 7.2.2. Analysis of Efficacy Analysis

See sections  $2\sim5$ .

<sup>\*</sup> estimated from ARISTOTLE and CER studies

<sup>\*\*</sup> averages of incidence rates shown in the Tables above

<sup>\*\*\*</sup> Calculated using an on-line calculator (Sample Size Survival Analysis (quesgen.com))

7.2.3. Summary of Analyses

Efficacy and safety analyses excluding descriptive summaries will be shown in the following table.

# 1) Unbalanced cohorts

| Outcome | Analysis Set | Supports Protocol<br>Objective Number | Subgroups | Statistical Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| The incidence rates of<br>stroke/SE and major<br>bleeding per 1,000<br>person-years | Unbalanced patients With high bleeding risk cohort vs without high bleeding risk cohort | NA | NA | 1000 person-years<br>(no statistical comparison) | Refer to 5.4 | No<br>imputation |
| Interaction analysis | Unbalanced patients With high bleeding risk cohort vs without high bleeding risk cohort | NA | NA | Cox proportional hazards model | With/without high<br>bleeding risk,<br>Warfarin/apixaban | No<br>imputation |

# 2) Balanced cohorts

| Outcome | Analysis Set | Supports Protocol<br>Objective Number | Subgroups | Statistical Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| Major bleeding | Balanced patients Warfarin vs. apixaban Cohorts | safety, primary | Whole cohort, primary analysis | Cox proportional hazards model | Refer to 5.4 | No<br>imputation |
| Major bleeding | Balanced patients Warfarin vs. apixaban Cohorts | safety, primary | Whole cohort, primary analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Major bleeding | Balanced patients Warfarin vs. apixaban Cohorts | safety, primary | Whole cohort, primary analysis | Incidence rate (per 1000 patient-year) | | No imputation |
| Major intracranial bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Cox proportional hazards model | Refer to 5.4 | No imputation |
| Major intracranial bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Major intracranial bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Incidence rate (per 1000 patient-year) | | No imputation |
| Major GI bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Cox proportional hazards model | Refer to 5.4 | No<br>imputation |
| Major GI bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Major GI bleeding | Balanced patients Warfarin vs. apixaban Cohorts | Safety<br>Secondary | Whole cohort, secondary analysis | Incidence rate (per 1000 patient-year) | | No<br>imputation |

| Outcome | Analysis Set | Supports Protocol<br>Objective Number | Subgroups | Statistical Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| Stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Primary | Whole cohort, secondary analysis | Cox proportional hazards model | Refer to 5.4 | No imputation |
| Stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Primary | Whole cohort, secondary analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Primary | Whole cohort, secondary analysis | Incidence rate (per 1000 patient-year) | | No imputation |
| Stroke | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Cox proportional hazards model | Refer to 5.4 | No imputation |
| Stroke | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Stroke | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Incidence rate (per 1000 patient-year) | | No imputation |
| SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Cox proportional hazards model | Refer to 5.4 | No imputation |
| SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| SE | Balanced patients Warfarin vs. apixaban Cohorts | Effectiveness<br>Secondary | Whole cohort, secondary analysis | Incidence rate (per 1000 patient-year) | | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Hypertension subgroup, exploratory analysis | 1000 person-years | Refer to 5.4 | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Hypertension subgroup, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Hypertension subgroup, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Liver dysfunction<br>subgroup, exprolatory<br>analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Liver dysfunction<br>subgroup, exprolatory<br>analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Liver dysfunction<br>subgroup, exprolatory<br>analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Renal impairment, exploratory analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Renal impairment, exploratory analysis | Incidence rate (per 100 patient-year) | | No imputation |

| Outcome | Analysis Set | Supports Protocol<br>Objective Number | Subgroups | Statistical Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| | | | | (no statistical comparison) | | |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Renal impairment Renal impairment, exprolatory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Bleeding history<br>subgroup, exploratory<br>analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Bleeding history<br>subgroup, exploratory<br>analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | <b>Balanced patients</b><br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Bleeding history<br>subgroup, exploratory<br>analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Concomitant use of antiplatelet drug, exploratory analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Concomitant use of antiplatelet drug, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Concomitant use of antiplatelet drug, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Age ✓ >80 y ✓ >90 y exploratory analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Age ✓ >80 y ✓ >90 y exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Age ✓ >80 y ✓ >90 y exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Peptic ulcer, exploratory analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |

| Outcome | Analysis Set | Supports Protocol<br>Objective Number | Subgroups | Statistical Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Peptic ulcer, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Peptic ulcer, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Active cancer, exploratory analysis | 1000 person-years | Refer to 5.4 | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Active cancer, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Active cancer, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Low body weight, exploratory analysis | 1000 person-years | Refer to 5.4 | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Low body weight, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Low body weight, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Diabetes mellitus, exploratory analysis | 1000 person-years | Refer to 5.4 | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Diabetes mellitus, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Diabetes mellitus, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Polypharmacy, exploratory analysis | 1000 person-years | Refer to 5.4 | No imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients<br>Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Polypharmacy, exploratory analysis | Incidence rate (per 100 patient-year) (no statistical comparison) | | No<br>imputation |
| Safety: Major Bleeding<br>Effectiveness: stroke/SE | Balanced patients Warfarin vs. apixaban Cohorts | Safety/effectiveness<br>Exploratory | Polypharmacy, exploratory analysis | Plot of Kaplan-Meier<br>Estimates | | No<br>imputation |

#### 8. LIST OF TABLES AND TABLE SHELLS

#### 9. REFERENCES

- 1. Lip GYH, Brechin CM, Lane DA. The global burden of atrial fibrillation and stroke: a systematic review of the epidemiology of atrial fibrillation in regions outside North America and Europe. Chest 2012;142:1489-1498.
- 2. Tomita F, Kohya T, Sakurai M, Kaji T, Yokoshiki H, Sato M, et al. Prevalence and clinical characteristics of patients with atrial fibrillation: analysis of 20,000 cases in Japan. Jpn Circ J 2000;64:653-658.
- 3. Kopecky SL, Gersh BJ, McGoon MD, Whisnant JP, Holmes DR, Jr., Ilstrup DM, et al. The natural history of lone atrial fibrillation. A population-based study over three decades. N Engl J Med 1987;317:669-674.
- 4. Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med 2009;361:1139-1151.
- 5. Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med 2011;365:981-992.
- 6. Kohsaka S, Murata T, Izumi N, Katada J, Wang F, Terayama Y. Bleeding risk of apixaban, dabigatran, and low-dose rivaroxaban compared with warfarin in Japanese patients with non-valvular atrial fibrillation: a propensity matched analysis of administrative claims data. Curr Med Res Opin 2017;33:1955-1963.
- 7. Kohsaka S, Katada J, Saito K, Terayama Y. Safety and effectiveness of apixaban in comparison to warfarin in patients with nonvalvular atrial fibrillation: a propensity-matched analysis from Japanese administrative claims data. Curr Med Res Opin 2018;34(9):1627-1634.
- 8. Kohsaka S, Katada J, Saito K, Jenkins A, Li B, Mardekian J, Terayama Y. Safety and effectiveness of non-vitamin K oral anticoagulants versus warfarin in real-world patients with non-valvular atrial fibrillation: a retrospective analysis of contemporary Japanese administrative claims data. Open Heart 2020 Apr 1;7(1):e001232.
- 9. Xu S, Ross C, Raebel MA, Shetterly S, Blanchette C, Smith D. Use of stabilized inverse propensity scores as weights to directly estimate relative risk and its confidence intervals. Value Health 2010;13:273-277
- 10. VanderWeele TJ and Ding P. Sensitivity Analysis in Observational Research: Introducing the E-Value. Ann Intern Med. 2017 Aug 15;167(4):268-274.

#### 10. APPENDICES

#### 10.1. APPENDIX 1: DATA DERIVATION DETAILS

Not applicable

# 10.2. APPENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS

Not applicable

# 10.3. APPENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY

# 10.3.1. List of diagnosis code

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| Atrial fibrillation | I48 | on 2 mm 2 m monor |
| Post-operative atrial fibrillation | 8847772 | Standard disease code |
| Valvular atrial fibrillation | 8846941 | Standard disease code |
| Rheumatic atrial fibrillation | I05 | |
| | 106 | |
| | I07 | |
| | I08 | |
| | 109 | |
| Mechanical-valvular atrial fibrillation | T820 | |
| Hyperthyroidism or thyrotoxicosis | E05 | |
| Heart failure | I110 | |
| | I500 | |
| | I501 | Exclude cardiac asthma |
| | I509 | |
| Hypertension | H208 | Include only hypertensive iridocyclitis |
| | H350 | Include only hypertensive retinopathy and hypertensive neuroretinopathy |
| | I10 | |
| | I110 | |
| | I119 | |
| | I120 | |
| | I129 | Include only hypertensive renal disease, hypertensive nephropathy and hypertensive nephrosclerosis |
| | I139 | |

| II50 | Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|---|
| TIS2 | • | | |
| TIS8 | | I151 | |
| Tis9 | | I152 | |
| Include only hypertensive intracerebral hemorrhage | | I158 | |
| Tital Hamour Hamour | | I159 | |
| Diabetes | | I619 | Include only hypertensive intracerebral hemorrhage |
| E11 | | I674 | |
| E12 | Diabetes | E10 | |
| E13 | | E11 | |
| E14 | | E12 | |
| Hemorrhage stroke | | E13 | |
| TIA | | E14 | |
| I62 | Hemorrhage stroke | I60 | |
| Ischemic stroke | | I61 | |
| 3489032 standard disease code | | I62 | Exclude non-traumatic extradural haemorrhage |
| 4371003 4379014 3448002 3448028 3489029 3489035 4379006 TIA | Ischemic stroke | I63 | |
| 4379014 3448002 3448028 3489029 3489035 4379006 | | 3489032 | standard disease code |
| | | 4371003 | - |
| 3448028 3489029 3489035 4379006 TIA | | 4379014 | - |
| 3489029 3489035 4379006 TIA | | 3448002 | 1 |
| | | 3448028 | 1 |
| $\begin{array}{c c} & & & \\ \hline \text{TIA} & & & \\ \hline & & & \\ \hline $ | | 3489029 | 1 |
| $\begin{array}{c c} TIA & H340 \\ \hline G450 \\ \hline G451 \\ \hline G458 \\ \hline G459 \\ \hline \\ Systemic embolism & I740 & Include only abdominal aortic embolism \\ \hline I741 & Include only aortic embolism \\ \hline \end{array}$ | | 3489035 | 1 |
| G450 G451 G458 G459 Systemic embolism I740 Include only abdominal aortic embolism I741 Include only aortic embolism | | 4379006 | 1 |
| G451 G458 G459 Systemic embolism I740 Include only abdominal aortic embolism I741 Include only aortic embolism | TIA | H340 | |
| G458 G459 Systemic embolism I740 Include only abdominal aortic embolism I741 Include only aortic embolism | | G450 | |
| G459 Systemic embolism I740 Include only abdominal aortic embolism I741 Include only aortic embolism | | G451 | |
| Systemic embolism I740 Include only abdominal aortic embolism I741 Include only aortic embolism | | G458 | |
| I741 Include only aortic embolism | | G459 | |
| · | Systemic embolism | I740 | Include only abdominal aortic embolism |
| 1 | | I741 | Include only aortic embolism |
| Include only acute arterial occlusive disease of arteries of upper extremities | | I742 | |
| Include only femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities | | 1743 | Include only femoral arterial occlusion and acute arterial |
| I744 | | I744 | |
| I745 Include only iliac artery embolism | | I745 | Include only iliac artery embolism |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| | I748 | Include only hepatic artery embolism |
| | I749 | Include only thromboembolism, embolic infarction, aortic embolism |
| Peripheral vascular disorder | 1702 | Include only atherosclerosis and arteriosclerosis obliterans |
| | 1709 | |
| | I731 | Include only Buerger's disease |
| | I739 | Exclude peripheral circulatory failure, cerebrovascular spasm, and angiospasm pf the extremities |
| | I742 | opacin, and angrospacin pr me sintenness |
| | I743 | |
| | I745 | |
| | I748 | Include only subclavian artery stenosis |
| Aortic plaque | 4400011 | Standard disease code |
| | 8837393 | Standard disease code |
| Coronary artery disease | 1200 | |
| | I201 | |
| | I208 | |
| | I209 | |
| | I210 | |
| | I211 | |
| | I212 | |
| | I213 | |
| | I214 | |
| | I240 | |
| | I241 | |
| | I248 | |
| | I251 | |
| | I252 | Exclude calcification of coronary artery |
| | I255 | |
| | I258 | Exclude coronary arteritis |
| | 1259 | |
| Myocardial infarction | 1200 | Exclude intermediate angina syndrome, preinfarction syndrome, initial arbeits angina, intermediate coronary syndrome |
| | I210 | |
| | I211 | |
| | I212 | |
| | I214 | |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| | I240 | |
| | I241 | Exclude Dressler syndrome |
| Renal impairment | I120 | |
| | I129 | |
| | I139 | |
| | N003 | |
| | N009 | |
| | N032 | |
| | N033 | |
| | N039 | |
| | N040 | |
| | N044 | |
| | N049 | |
| | N052 | |
| | N055 | |
| | N058 | |
| | N059 | |
| | N170 | |
| | N171 | |
| | N172 | |
| | N178 | |
| | N179 | |
| | N189 | |
| | N19 | Exclude renal anemia, afunctional kidney, and alimentary proteinuria |
| Liver dysfunction | B150 | |
| | B159 | |
| | B162 | |
| | B169 | |
| | B171 | |
| | B172 | |
| | B178 | |
| | B179 | |
| | B181 | |
| | B182 | |
| | B189 | |
| | B190 | |
| | B199 | |

| C220 K700 K701 K703 K709 K716 K720 K721 K729 K730 K732 K738 K738 K739 K744 K741 K743 K744 K745 K746 K750 K751 K750 K751 K750 K761 K762 K763 K766 K767 K768 K769 C01 C02 C03 C04 C04 C04 C05 C06 C07 C07 C07 C08 C08 C09 C00 C01 C02 C03 C04 C00 C01 C02 C03 C04 C00 C01 C02 C03 C04 C00 C01 C02 C03 C04 C00 C01 C02 C03 C04 C06 C07 C07 C08 C09 C00 C01 C02 C03 C04 C06 C07 C08 C09 C09 C00 C00 | Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|---|
| K701 | | | |
| K703 K709 K716 K720 K721 K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C03 C04 | | K700 | |
| K709 K716 K720 K721 K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 | | K701 | |
| K716 K720 K721 K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K752 K760 K761 K762 K763 K766 K767 K768 K769 Cancer | | K703 | |
| K720 K721 K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K709 | |
| K721 K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K716 | |
| K729 K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K720 | |
| K730 K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K721 | |
| K732 K738 K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K729 | |
| K738 K739 K740 K741 K743 K744 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer Cancer Coo Cool | | K730 | |
| K739 K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K732 | |
| K740 K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer Col C01 C02 C03 C04 | | K738 | |
| K741 K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 C05 C04 C05 C06 C0 | | K739 | |
| K743 K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 C05 C06 C06 | | K740 | |
| K744 K745 K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 C04 C04 C04 C04 C04 C04 C05 C04 C06 C07 C07 C07 C08 C09 | | K741 | |
| K745 K746 K750 K751 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K768 Cancer Coo Coo Coo Coo Coo Coo Coo C | | K743 | |
| K746 K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K744 | |
| K750 K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer Coo Coo Coo Coo Coo Coo Coo C | | K745 | |
| K751 K754 K759 K760 K761 K762 K763 K766 K767 K768 K768 K769 Cancer C00 C01 C02 C03 C04 | | K746 | |
| K754 K759 K760 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K750 | |
| K759 K760 K761 K761 K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 C04 C04 C04 C04 C04 C04 C05 C06 C06 C06 C06 C06 C07 C07 | | K751 | |
| K760 | | K754 | |
| K761 K762 K763 K766 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 C04 C04 C04 C04 C04 C04 C05 C06 C06 C06 C07 C07 C08 C09 | | K759 | |
| K762 K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K760 | |
| K763 K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K761 | |
| K766 K767 K768 K769 Cancer C00 C01 C02 C03 C04 | | K762 | |
| K767 | | K763 | |
| K768 K769 Cancer C00 C01 C02 C03 C04 | | K766 | |
| K769 Cancer C00 C01 C02 C03 C04 C04 C04 C04 C04 C05 C06 C07 C08 C08 C08 C08 C08 C08 C09 | | K767 | |
| Cancer C00 C01 C02 C03 C04 | | K768 | |
| C01<br>C02<br>C03<br>C04 | | K769 | |
| C02<br>C03<br>C04 | Cancer | C00 | |
| C03<br>C04 | | C01 | |
| C04 | | C02 | |
| | | C03 | |
| | | C04 | |
| | | C05 | |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| V | C06 | |
| | C07 | |
| | C08 | |
| | C09 | |
| | C10 | |
| | C11 | |
| | C12 | |
| | C13 | |
| | C14 | |
| | C15 | |
| | C16 | |
| | C17 | |
| | C18 | |
| | C19 | |
| | C20 | |
| | C21 | |
| | C22 | |
| | C23 | |
| | C24 | |
| | C25 | |
| | C26 | |
| | C30 | |
| | C31 | |
| | C32 | |
| | C33 | |
| | C34 | |
| | C37 | |
| | C38 | |
| | C40 | |
| | C41 | |
| | C43 | |
| | C44 | |
| | C45 | |
| | C46 | |
| | C47 | |
| | C48 | |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| · | C49 | |
| | C50 | |
| | C51 | |
| | C52 | |
| | C53 | |
| | C54 | |
| | C55 | |
| | C56 | |
| | C57 | |
| | C58 | |
| | C60 | |
| | C61 | |
| | C62 | |
| | C63 | |
| | C64 | |
| | C65 | |
| | C66 | |
| | C67 | |
| | C68 | |
| | C69 | |
| | C70 | |
| | C71 | |
| | C72 | |
| | C73 | |
| | C74 | |
| | C75 | |
| | C76 | |
| | C78 | |
| | C79 | |
| | C80 | |
| | C81 | |
| | C82 | |
| | C83 | |
| | C84 | |
| | C85 | |
| | C88 | |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| | C90 | |
| | C91 | |
| | C92 | |
| | C93 | |
| | C94 | |
| | C95 | |
| | C96 | |
| | C97 | |
| | D00 | |
| | D01 | |
| | D02 | |
| | D03 | |
| | D04 | |
| | D05 | |
| | D06 | |
| | D07 | |
| | D09 | |
| | D10 | |
| | D11 | |
| | D12 | |
| | D13 | |
| | D14 | |
| | D15 | |
| | D16 | |
| | D17 | |
| | D18 | |
| | D19 | |
| | D20 | |
| | D21 | |
| | D22 | |
| | D23 | |
| | D24 | |
| | D25 | |
| | D27 | |
| | D28 | |
| | D29 | |

| Variable Used<br>in Study | ICD-10<br>Code* | Additional rules<br>on Data Extraction |
|---|---|---|
| • | D30 | |
| | D31 | |
| | D32 | |
| | D33 | |
| | D34 | |
| | D35 | |
| | D36 | |
| | D37 | |
| | D38 | |
| | D39 | |
| | D40 | |
| | D41 | |
| | D42 | |
| | D43 | |
| | D44 | |
| | D45 | |
| | D46 | |
| | D48 | |

# 10.3.2. List of procedure code

| Procedure | Procedure Code |
|-----------------|----------------|
| Cardiac surgery | 150138210 |
| | 150138310 |
| | 150138410 |
| | 150138510 |
| | 150359210 |
| | 150138710 |
| | 150140510 |
| | 150140610 |
| | 150140710 |
| | 150139010 |
| | 150140810 |
| | 150318010 |
| | 150317810 |
| | 150318110 |
| | 150331450 |

| 150331550 150331950 150332050 150317910 150318210 150140010 150139210 150139910 150374910 150374910 150375110 150260350 150284310 150359310 150363310 150375210 150375210 150375310 150375310 150375310 150375410 160107550 150139810 150318310 150318310 150318310 150318310 150318310 150318310 150318310 150318510 150318510 | Procedure | Procedure Code |
|---|---|---|
| 150332050 150317910 150318210 150140010 150139210 150153910 150375010 150375010 150375110 150260350 150284310 150359310 150359310 150359310 150375210 150375210 150375210 150375310 150375210 150375310 150375410 160107550 150139810 150145810 150145710 150145810 150145710 150146010 150318410 150318510 150318510 150318510 150318510 15032770 150143110 150331650 150332150 150332150 150331710 150318710 150319310 | | 150331550 |
| 150317910 150318210 150140010 150139210 150153910 150375910 150375010 150375110 150260350 150284310 150359310 150375210 150375210 150375210 150375310 150375310 150375310 150375410 160107550 150139810 150139810 150145710 150145710 150145810 150145910 150145910 150318410 150318510 150318510 150332770 150143010 15031810 150332150 150332150 150332150 150331910 150319310 | | 150331950 |
| 150318210 150140010 150139210 150153910 150375010 150375010 150375110 150260350 150284310 150359310 150363310 150375210 150375210 150375210 150375310 150375310 150375410 160107550 150139810 150139810 150139810 150145710 150145710 150145810 150145910 150146010 150318410 150318410 150302770 150143010 150143110 150331650 150332150 150318710 150319310 150318810 | | 150332050 |
| 150140010 150139210 150133910 150374910 150375110 150260350 150284310 150263310 150375210 150375210 150375310 150375310 150375310 150375310 150375310 150375410 160107550 150139810 150139810 150145710 150145710 150145810 150145810 150145810 150145910 150318310 150318310 150318510 150318510 150318510 150318510 150318510 150318710 150318710 150318710 150318710 150319310 150319310 150319310 150319310 150319310 150318810 | | 150317910 |
| 150139210 150153910 150374910 150375010 150375010 15026350 15026350 150263510 150263310 150375210 150375210 150375210 150375310 150375310 150375410 160107550 150139810 150139810 150145710 150145710 150145810 150145810 150145810 150145910 150318310 150318310 150145910 150318310 150145910 150318310 150145910 150318510 150318510 150318510 150318510 15033150 15033150 15033150 15033150 15033150 15033150 150318710 150319310 150319310 | | 150318210 |
| 150153910 150374910 150375010 150375110 150260350 150284310 150359310 150375210 150375210 150375210 150375310 150375410 160107550 150139810 150318310 150145710 150145810 150145910 150145910 150145910 150145910 150318410 150318510 150302770 150143010 150332150 150332150 150332150 150318710 | | 150140010 |
| 150374910 150375010 150375110 150260350 150284310 150359310 150263310 150375210 150375210 150375310 150375410 160107550 150139810 150139810 150139910 150318310 150145710 150145710 150145810 150145810 150145910 150146010 150318410 150318510 150302770 150143010 150143110 150332150 150332150 150318710 150319010 150319310 150319310 150318810 | | 150139210 |
| 150375010 150375110 150260350 150284310 150359310 150263310 150263310 150375210 150375310 150375410 160107550 150139810 150139910 150318310 150145710 150145710 150145810 150145910 150145910 150318410 150318510 150302770 150143010 150331650 150332150 150332150 150318710 150319010 150319310 150319310 | | 150153910 |
| 150375110 150260350 150284310 150359310 150263310 150375210 150375210 150375310 150375410 160107550 150139810 150318310 150318310 150145710 150145710 150145810 150145910 150318410 150318510 | | 150374910 |
| 150260350 150284310 150359310 150263310 150375210 150375210 150375310 160107550 150139810 150318310 150318310 150145710 150145810 150145810 150145910 150318410 150318410 150318510 150318510 150318510 15032770 150143010 150331650 150332150 1503318710 150319010 150318810 | | 150375010 |
| 150284310 150359310 150263310 150375210 150375310 150375410 160107550 150139810 150318310 150318310 150145710 150145710 150145810 150145910 150318410 150318410 150318510 150302770 150143010 150143110 150331650 150332150 150318710 150318710 150318810 | | 150375110 |
| 150359310 150263310 150375210 150375310 150375410 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150318410 150318510 150318510 150302770 150143010 150331650 150332150 150318710 150319310 150319310 | | 150260350 |
| 150263310 150375210 150375310 150375410 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150146010 150318410 150318510 15032770 150143010 150143110 150331650 150332150 150319310 150319310 150319310 | | 150284310 |
| 150375210 150375310 150375410 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150146010 150318410 150318510 150318510 150302770 150143010 150331650 150332150 150332150 150318710 150319310 150318810 | | 150359310 |
| 150375310 150375410 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150318410 150318410 150318510 150302770 150143010 150331650 150332150 150318710 150319010 150319310 150318810 | | 150263310 |
| 150375410 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150318410 150318410 150318510 150302770 150143010 150331650 150332150 150318710 150319010 150319310 | | 150375210 |
| 160107550 150139810 150139910 150318310 150145710 150145810 150145910 150146010 150318410 150318510 150302770 150143010 150143110 150331650 150332150 150318710 150319310 150318810 | | 150375310 |
| 150139810 150139910 150318310 150145710 150145810 150145910 150146010 150318410 150318510 150302770 150143010 150331650 150332150 150318710 150319310 150319310 | | 150375410 |
| 150139910 150318310 150145710 150145810 150145910 150146010 150318410 150318510 150302770 150143010 150143110 150331650 150332150 150318710 150319310 150318810 | | 160107550 |
| 150318310 150145710 150145810 150145910 150318410 150318410 150318510 150302770 150143010 150331650 150332150 150318710 150319010 150318810 | | 150139810 |
| 150145710 150145810 150145910 150146010 150318410 150318510 150302770 150143010 150143110 150331650 150332150 150318710 150319010 150319310 150318810 | | 150139910 |
| 150145810<br>150146010<br>150318410<br>150318510<br>150302770<br>150143010<br>150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150318810 | | 150318310 |
| 150145910 150146010 150318410 150318510 150302770 150143010 150143110 150331650 150332150 150318710 150319010 150319310 150318810 | | 150145710 |
| 150146010 150318410 150318510 150302770 150143010 150331650 150332150 150318710 150319310 150318810 | | 150145810 |
| 150318410<br>150318510<br>150302770<br>150143010<br>150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150319010 | | 150145910 |
| 150318510<br>150302770<br>150143010<br>150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150319310 | | 150146010 |
| 150302770<br>150143010<br>150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150319310 | | 150318410 |
| 150143010<br>150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150319310<br>150318810 | | 150318510 |
| 150143110<br>150331650<br>150332150<br>150318710<br>150319010<br>150319310 | | 150302770 |
| 150331650<br>150332150<br>150318710<br>150319010<br>150319310<br>150318810 | | 150143010 |
| 150332150<br>150318710<br>150319010<br>150319310<br>150318810 | | 150143110 |
| 150318710<br>150319010<br>150319310<br>150318810 | | |
| 150319010<br>150319310<br>150318810 | | 150332150 |
| 150319310<br>150318810 | | 150318710 |
| 150318810 | | 150319010 |
| | | 150319310 |
| 150319110 | | 150319110 |
| Procedure | Procedure Code |
|-----------|----------------|
| | 150319410 |
| | 150328750 |
| | 150328850 |
| | 150331750 |
| | 150331850 |
| | 150332250 |
| | 150332350 |
| | 150318910 |
| | 150319210 |
| | 150319510 |
| | 150318610 |
| | 150141010 |
| | 150279510 |
| | 150279610 |
| | 150141410 |
| | 150141610 |
| | 150369950 |
| | 150141710 |
| | 150359470 |
| | 150143610 |
| | 150260050 |
| | 150143710 |
| | 150143810 |
| | 150141510 |
| | 150375570 |
| | 150375670 |
| | 150375770 |
| | 150319610 |
| | 150292910 |
| | 150139310 |
| | 150140910 |
| | 150242550 |
| | 150244910 |
| | 150245010 |
| | 150359510 |
| | 150359610 |
| | 150381150 |
| | 150381250 |

| 150381350<br>150381450<br>150150010<br>150381550<br>150275910<br>150359710<br>150359810<br>150359910 |
|---|
| 150150010<br>150381550<br>150275910<br>150359710<br>150359810 |
| 150381550<br>150275910<br>150359710<br>150359810 |
| 150275910<br>150359710<br>150359810 |
| 150359710<br>150359810 |
| 150359810 |
| 150359910 |
| 130337710 |
| 150381650 |
| 150381750 |
| 150381850 |
| 150381950 |
| 150150110 |
| 150382050 |
| 150245110 |
| 150245210 |
| 150375870 |
| 150375970 |
| 150376070 |
| 150141210 |
| 150301310 |
| 150267850 |
| 150319710 |
| 150151810 |
| 150376110 |
| 150139110 |
| 150319810 |
| 150138810 |
| 150151910 |
| 150320010 |
| 150346410 |
| 150320110 |
| 150147150 |
| 150144110 |
| 150320210 |
| 150320310 |
| 150142710 |
| 150139410 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150320410 |
| | 150142910 |
| | 150320510 |
| | 150260150 |
| | 150346510 |
| | 150145110 |
| | 150145010 |
| | 150376210 |
| | 150376310 |
| | 150143250 |
| | 150143350 |
| | 150143450 |
| | 150143550 |
| | 150283250 |
| | 150283350 |
| | 150283450 |
| | 150283550 |
| | 150144910 |
| | 150139610 |
| | 150142410 |
| | 150141810 |
| | 150141910 |
| | 150320610 |
| | 150142050 |
| | 150142110 |
| | 150142210 |
| | 150142310 |
| | 150142810 |
| | 150144010 |
| | 150320710 |
| | 150144210 |
| | 150144550 |
| | 150147410 |
| | 150147510 |
| | 150320810 |
| | 150320910 |
| | 150144410 |
| | 150144650 |

| 150144750 150146510 150146610 150321010 150321110 150321210 150376470 150146810 150321310 15014510 150321310 150145210 15032910 150329810 150145310 150329910 150330010 150147010 150330110 150330310 1503303270 150145410 150145410 | Procedure | Procedure Code |
|---|---|---|
| 150146610 150321010 15032110 150321210 150376470 150146910 150146810 150321310 150142510 150329810 150143510 150329910 150139510 150330010 150330010 150330110 150330110 150321510 15032150 150147310 150321510 150321710 150321710 150330310 | | 150144750 |
| 15032100 15032110 15032110 150376470 150146910 150146810 150142510 150329810 150142510 150329810 150139510 150339910 150139510 150330010 150147010 150330110 150321410 150321410 150321410 150321410 15032160 150321410 15032160 150321410 150321710 150321810 150321710 150321710 15033010 15033010 15033010 15032770 15032170 150330310 150376770 150330310 150376770 150293010 150330410 150330410 150330410 | | 150146510 |
| 150321110 150321210 150376470 150146910 150146810 150321310 150142510 150142510 1501329810 150145310 150139510 150139510 150139510 150330010 150147010 150330110 150321410 150321410 150321410 150321510 150376670 150147310 15014650 150141310 150321810 150321810 150321910 150321910 150316710 150321710 150330310 150330310 150330310 150376770 150293010 150302870 | | 150146610 |
| 150321210 150376470 150146910 150146810 150142510 150329810 150329810 150329910 150339010 150330010 150376570 150321510 150321510 150376670 150147310 1503150 150321610 150321610 150321610 150321610 150321610 150321710 150321710 150330110 1503276770 15032010 150330310 150376770 150300410 150302870 | | 150321010 |
| 150376470 150146910 150146810 150321310 150329810 150329910 150339910 150339910 150330010 150330010 150330110 150330110 150330110 150330110 15033110 150321410 150321510 150376670 150147310 150147310 150145650 150141310 150321810 150321810 150321910 150330310 150321710 150330310 150376770 150293010 150330410 150302870 | | 150321110 |
| 150146910 150146810 150321310 150329810 150142510 150329910 150339910 150339910 150330010 150147010 150330110 150321410 150321410 150321510 150376670 150147310 150147310 15034650 150147310 150321810 150321810 150321810 150321810 150321910 150321910 150321710 150330310 150330310 150330310 150330310 150330410 150330410 150302870 | | 150321210 |
| 150146810 150321310 150142510 150329810 150145310 150329910 150139510 150330010 150147010 150330110 150330110 15033670 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321810 150321910 150321910 150321710 150321710 150330210 150330310 150330310 150330310 150330310 150330410 150302870 | | 150376470 |
| 150321310 150142510 150329810 150145310 150329910 150139510 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150147310 15014550 150141310 150321610 150321610 150321710 15033010 150330210 150330310 150330310 150330310 150330410 150302870 | | 150146910 |
| 150142510 150329810 150145310 150329910 150139510 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150147310 150145650 150141310 150321810 150321810 150321910 150321910 150321910 150321910 150321710 150321710 150330110 15030310 15030310 150303010 15030410 150302870 | | 150146810 |
| 150329810 150145310 150329910 150139510 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321910 150321910 150321710 150321710 15033010 15033010 15033010 150330310 150330410 150302870 | | 150321310 |
| 150145310 150329910 150139510 150330010 150147010 150330110 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321910 150321710 150330110 150330110 150330110 150330310 150376770 150293010 1503045510 150145510 | | 150142510 |
| 150329910 150139510 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321910 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150302870 | | 150329810 |
| 150139510 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150147310 150145650 150141310 150321810 150321810 150321610 150321710 150330310 150330310 150330310 150330410 15033045510 150145510 150302870 | | 150145310 |
| 150330010 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321610 150321910 150321710 150330110 150330110 150330310 150376770 150293010 150330410 150302870 | | 150329910 |
| 150147010 150330110 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321910 150321910 150321710 150330210 150330310 150330310 150330410 150330410 150145510 150302870 | | 150139510 |
| 150330110 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321810 150321910 150321910 150321710 150330210 150330310 150330310 150376770 150293010 150330410 150145510 150302870 | | 150330010 |
| 150376570 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321610 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150302870 | | 150147010 |
| 150321410 150321510 150376670 150147310 150145650 150141310 150321810 150321610 150321910 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150145510 150302870 | | 150330110 |
| 150321510 150376670 150147310 150145650 150141310 150321810 150321610 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150302870 | | 150376570 |
| 150376670 150147310 150145650 150141310 150321810 150321610 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150145510 150302870 | | 150321410 |
| 150147310<br>150145650<br>150141310<br>150321810<br>150321610<br>150321910<br>150146710<br>150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150321510 |
| 150145650 150141310 150321810 150321610 150321910 150146710 150321710 150330210 150330310 150376770 150293010 150330410 150145510 150302870 | | 150376670 |
| 150141310 150321810 150321610 150321910 150321710 150330210 150330310 150376770 150293010 150330410 150145510 150302870 | | 150147310 |
| 150321810<br>150321610<br>150321910<br>150146710<br>150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150145650 |
| 150321610<br>150321910<br>150146710<br>150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150141310 |
| 150321910<br>150146710<br>150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150321810 |
| 150146710<br>150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150321610 |
| 150321710<br>150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150321910 |
| 150330210<br>150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150146710 |
| 150330310<br>150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150321710 |
| 150376770<br>150293010<br>150330410<br>150145510<br>150302870 | | 150330210 |
| 150293010<br>150330410<br>150145510<br>150302870 | | 150330310 |
| 150330410<br>150145510<br>150302870 | | 150376770 |
| 150145510<br>150302870 | | 150293010 |
| 150302870 | | 150330410 |
| | | 150145510 |
| 150145410 | | 150302870 |
| f I | | 150145410 |

| 150322010 150322110 150144310 150147250 150346610 150144810 150253810 150253910 150275610 150346710 150362810 150303310 150267310 150140110 | |
|---|---|
| 150144310<br>150147250<br>150346610<br>150144810<br>150253810<br>150253910<br>150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150147250 150346610 150144810 150253810 150253910 150275610 150346710 150262810 150303310 150267310 150140110 | |
| 150346610<br>150144810<br>150253810<br>150253910<br>150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150144810<br>150253810<br>150253910<br>150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150253810<br>150253910<br>150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150253910<br>150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150275610<br>150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150346710<br>150262810<br>150303310<br>150267310<br>150140110 | |
| 150262810<br>150303310<br>150267310<br>150140110 | |
| 150303310<br>150267310<br>150140110 | |
| 150267310<br>150140110 | _ |
| 150140110 | |
| | _ |
| 150140210 | _ |
| 150140410 | |
| 150346910 | |
| 150347010 | |
| 150303210 | |
| 150322210 | |
| 150275210 | |
| 150275310 | |
| 150336910 | |
| 150337010 | |
| 150360010 | |
| 150148010 | |
| 150148110 | |
| 150147610 | |
| 150147910 | |
| 150147770 | |
| 150147870 | |
| 150347170 | |
| 150275870 | |
| 150262910 | |
| 150275710 | |
| 150266110 | |
| 150382650 | |
| 150266210 | |

| Procedure | Procedure Code |
|---------------------------------------------|----------------|
| | 150382750 |
| | 150301810 |
| | 150382850 |
| | 150303410 |
| | 150303510 |
| | 150360110 |
| | 150360210 |
| | 150360310 |
| | 150360410 |
| | 150303610 |
| | 150303710 |
| | 150322410 |
| | 150322610 |
| Ablation | 150346710 |
| | 150262810 |
| | 150303310 |
| | 150346870 |
| | 150370050 |
| Electrical defibrillation | 140051410 |
| | 140010310 |
| | 140055010 |
| | 150275210 |
| | 150275310 |
| | 150336910 |
| | 150337010 |
| | 150370550 |
| Heart valve prosthesis implantation surgery | 150141410 |
| | 150141610 |
| | 150141710 |
| | 150359470 |
| | 150369950 |
| | 150331950 |
| | 150332050 |
| | 150332150 |
| | 150328850 |
| | 150332250 |
| | 150332350 |
| | 150141510 |

| Procedure | Procedure Code |
|-----------|----------------|
| | 150375570 |
| | 150375670 |
| | 150375770 |
| | 150244910 |
| | 150359510 |
| | 150381150 |
| | 150381250 |
| | 150359710 |
| | 150359810 |
| | 150381650 |
| | 150381750 |
| | 150283450 |

## 10.3.3. Effectiveness endpoints

| Disease | ICD10<br>code | Standard<br>disease code | Note |
|---|---|---|---|
| Поточиводо | I60 | | |
| Hemorrhage<br>stroke | I61 | | |
| Stroke | I62 | | Exclude non-traumatic extradural haemorrhage |
| | I63 | | |
| | | 3489032 | |
| | | 4371003 | |
| | | 4379014 | |
| Ischemic stroke | | 3448002 | |
| | | 3448028 | |
| | | 3489029 | |
| | | 3489035 | |
| | | 4379006 | |
| | H340 | | |
| | G450 | | |
| TIA | G451 | | |
| | G458 | | |
| | G459 | | |
| | I740 | | Include only abdominal aortic embolism |
| | I741 | | Include only aortic embolism |
| | I742 | | Include only acute arterial occlusive disease of arteries of upper extremities |
| Systemic | I743 | | Include only femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities |
| embolism | I744 | | |
| | I745 | | Include only iliac artery embolism |
| | I748 | | Include only hepatic artery embolism |
| | I749 | | Include only thromboembolism, embolic infarction, aortic embolism |

PFIZER CONFIDENTIAL

Disease ICD10 Standard Note

I748 Include only subclavian artery stenosis

## 10.3.4. Safety endopoints

| Disease | ICD10<br>code | Standard<br>disease code | Note |
|---|---|---|---|
| Major bleeding | | | Refer to 10.3.5 |
| | I600 | | Subarachnoid haemorrhage from carotid siphon and bifurcation |
| | I601 | | Subarachnoid haemorrhage from middle cerebral artery |
| | 1602 | | Subarachnoid haemorrhage from anterior communicating artery |
| | 1603 | | Subarachnoid haemorrhage from posterior communicating artery |
| | I604 | | Subarachnoid haemorrhage from basilar artery |
| | I605 | | Subarachnoid haemorrhage from vertebral artery |
| | I606 | | Subarachnoid haemorrhage from other intracranial arteries |
| | I607 | | Subarachnoid haemorrhage from intracranial artery, unspecified |
| | I608 | | Other subarachnoid haemorrhage |
| | I609 | | Subarachnoid haemorrhage, unspecified |
| | I610 | | Intracerebral haemorrhage in hemisphere, subcortical |
| Intracranial | I611 | | Intracerebral haemorrhage in hemisphere, cortical |
| bleeding | I613 | | Intracerebral haemorrhage in brain stem |
| | I614 | | Intracerebral haemorrhage in cerebellum |
| | I615 | | Intracerebral haemorrhage, intraventricular |
| | I616 | | Intracerebral haemorrhage, multiple localized |
| | I618 | | Other intracerebral haemorrhage |
| | I619 | | Intracerebral haemorrhage, unspecified |
| | I620 | | Subdural haemorrhage (acute)(nontraumatic) |
| | I621 | | Nontraumatic extradural haemorrhage |
| | I629 | | Intracranial haemorrhage (nontraumatic), unspecified |
| | I690 | | Sequelae of subarachnoid haemorrhage |
| | I691 | | Sequelae of intracerebral haemorrhage |
| | S064 | | Epidural haemorrhage |
| | S065 | | Traumatic subdural haemorrhage |
| | S066 | | Traumatic subarachnoid haemorrhage |
| | S068 | | Other intracranial injuries |
| | I850 | | Oesophageal varices with bleeding |
| | K226 | | Gastro-oesophageal laceration-haemorrhage syndrome |
| | K228 | | Other specified diseases of oesophagus |
| | K250 | | Acute with haemorrhage |
| GI bleeding | K252 | | Gastric ulcer, Acute with both haemorrhage and perforation |
| | K254 | | Gastric ulcer, Chronic or unspecified with haemorrhage |
| | K256 | | Gastric ulcer, Chronic or unspecified with both haemorrhage and perforation |
| | K260 | | Duodenal ulcer, Acute with haemorrhage |

| Disease | ICD10<br>code | Standard<br>disease code | Note |
|---|---|---|---|
| | K262 | | Duodenal ulcer, Acute with both haemorrhage and perforation |
| | K264 | | Duodenal ulcer, Chronic or unspecified with haemorrhage |
| | K266 | | Duodenal ulcer, Chronic or unspecified with both haemorrhage and perforation |
| | K270 | | Acute duodenal tumor with haemorrhage |
| | K284 | | Gastrojejunal ulcer, Chronic or unspecified with haemorrhage |
| | K290 | | Acute haemorrhagic gastritis |
| | K625 | | Haemorrhage of anus and rectum |
| | K920 | | Haematemesis |
| | K921 | | Melaena |
| | K922 | | Gastrointestinal haemorrhage, unspecified |

#### **10.3.5.** bleeding

Procedure for definition of "bleeding"

Step 1. To extract the following group A or group B from MDV data base.

Group A: ICD-10 name includes "出血 (bleeding)" or "血腫 (ecchymoma)"

Group B: Disease name includes "出血 (bleeding)" or "血腫 (ecchymoma)"

Step 2. To select disease names considered to be relevant to side effect of OAC individually from disease names excluded in Step 1.

Step 3. To exclude disease names which are not considered to be relevant to side effect of OAC from the disease names included in Step 1.

| ICD-10 | ICD10Name |
|---|---|
| A162 | Tuberculosis of lung, without mention of bacteriological or histological confirmation |
| A165 | Tuberculous pleurisy, without mention of bacteriological or histological confirmation |
| B303 | Acute epidemic haemorrhagic conjunctivitis (enteroviral) |
| D500 | Iron deficiency anaemia secondary to blood loss (chronic) |
| D62 | Acute post haemorrhagic anaemia |
| D66 | Hereditary factor VIII deficiency |
| D683 | Haemorrhagic disorder due to circulating anticoagulants |
| D698 | Other specified haemorrhagic conditions |
| D699 | Haemorrhagic condition, unspecified |
| E078 | Other specified disorders of thyroid |
| E274 | Other and unspecified adrenocortical insufficiency |
| G361 | Acute and subacute haemorrhagic leukoencephalitis [Hurst] |
| G951 | Vascular myelopathies |
| G968 | Other specified disorders of central nervous system |
| H052 | Exophthalmic conditions |
| H113 | Conjunctival haemorrhage |

| ICD-10 | ICD10Name |
|---|---|
| H168 | Other keratitis |
| H208 | Other iridocyclitis |
| H210 | Hyphaema |
| H313 | Choroidal haemorrhage and rupture |
| H350 | Background retinopathy and retinal vascular changes |
| H356 | Retinal haemorrhage |
| H357 | Separation of retinal layers |
| H405 | Glaucoma secondary to other eye disorders |
| H431 | Vitreous haemorrhage |
| H448 | Other disorders of globe |
| H470 | Disorders of optic nerve, not elsewhere classified |
| H603 | Other infective otitis externa |
| H669 | Otitis media, unspecified |
| H738 | Other specified disorders of tympanic membrane |
| H922 | Otorrhagia |
| I213 | Acute transmural myocardial infarction of unspecified site |
| I230 | Haemopericardium as current complication following acute myocardial infarction |
| I312 | Haemopericardium, not elsewhere classified |
| I600 | Subarachnoid haemorrhage from carotid siphon and bifurcation |
| I601 | Subarachnoid haemorrhage from middle cerebral artery |
| I602 | Subarachnoid haemorrhage from anterior communicating artery |
| I603 | Subarachnoid haemorrhage from posterior communicating artery |
| I604 | Subarachnoid haemorrhage from basilar artery |
| I605 | Subarachnoid haemorrhage from vertebral artery |
| I606 | Subarachnoid haemorrhage from other intracranial arteries |
| I607 | Subarachnoid haemorrhage from intracranial artery, unspecified |
| I608 | Other subarachnoid haemorrhage |
| I609 | Subarachnoid haemorrhage, unspecified |
| I610 | Intracerebral haemorrhage in hemisphere, subcortical |
| I611 | Intracerebral haemorrhage in hemisphere, cortical |
| I613 | Intracerebral haemorrhage in brain stem |
| I614 | Intracerebral haemorrhage in cerebellum |
| I615 | Intracerebral haemorrhage, intraventricular |
| I616 | Intracerebral haemorrhage, multiple localized |
| I618 | Other intracerebral haemorrhage |
| I619 | Intracerebral haemorrhage, unspecified |
| I620 | Subdural haemorrhage (acute)(nontraumatic) |
| I621 | Nontraumatic extradural haemorrhage |
| I629 | Intracranial haemorrhage (nontraumatic), unspecified |
| I638 | Other cerebral infarction |
| I690 | Sequelae of subarachnoid haemorrhage |
| I691 | Sequelae of intracerebral haemorrhage |

| ICD-10 | ICD10Name |
|---|---|
| I780 | Hereditary haemorrhagic telangiectasia |
| I788 | Other diseases of capillaries |
| I841 | Internal hemorrhoid with other complications |
| I844 | External hemorrhoid with other complications |
| I848 | Unspecified hemorrhoid with other complications |
| 1850 | Oesophageal varices with bleeding |
| I864 | Gastric varices |
| J041 | Acute tracheitis |
| J339 | Nasal polyp, unspecified |
| J90 | Pleural effusion, not elsewhere classified |
| J942 | Haemothorax |
| J950 | Tracheostomy malfunction |
| K049 | Other and unspecified diseases of pulp and periapical tissues |
| K068 | Other specified disorders of gingiva and edentulous alveolar ridge |
| K121 | Other forms of stomatitis |
| K137 | Other and unspecified lesions of oral mucosa |
| K148 | Other diseases of tongue |
| K226 | Gastro-oesophageal laceration-haemorrhage syndrome |
| K228 | Other specified diseases of oesophagus |
| K250 | Acute with haemorrhage |
| K252 | Gastric ulcer, Acute with both haemorrhage and perforation |
| K254 | Gastric ulcer, Chronic or unspecified with haemorrhage |
| K256 | Gastric ulcer, Chronic or unspecified with both haemorrhage and perforation |
| K260 | Duodenal ulcer, Acute with haemorrhage |
| K262 | Duodenal ulcer, Acute with both haemorrhage and perforation |
| K264 | Duodenal ulcer, Chronic or unspecified with haemorrhage |
| K266 | Duodenal ulcer, Chronic or unspecified with both haemorrhage and perforation |
| K270 | Acute duodenal tumor with haemorrhage |
| K284 | Gastrojejunal ulcer, Chronic or unspecified with haemorrhage |
| K290 | Acute haemorrhagic gastritis |
| K571 | Diverticular disease of small intestine without perforation or abscess |
| K573 | Diverticular disease of smart intestine without perforation of abscess Diverticular disease of large intestine without perforation or abscess |
| K625 | Haemorrhage of anus and rectum |
| K661 | Haemoperitoneum |
| K762 | Central haemorrhagic necrosis of liver |
| K768 | Other specified diseases of liver |
| K85 | Acute pancreatitis |
| K920 | Haematemesis |
| K921 | Melaena |
| K922 | Gastrointestinal haemorrhage, unspecified |
| L508 | Other urticaria |
| M250 | Haemarthrosis |
| | I . |

| ICD-10 | ICD10Name |
|---|---|
| N029 | Recurrent and persistent haematuria, Unspecified |
| N288 | Other specified disorders of kidney and ureter |
| N300 | Acute cystitis |
| N304 | Irradiation cystitis |
| N309 | Cystitis, unspecified |
| N328 | Other specified disorders of bladder |
| N368 | Other specified disorders of urethra |
| N421 | Congestion and haemorrhage of prostate |
| N488 | Other specified disorders of penis |
| N501 | Vascular disorders of male genital organs |
| N645 | Other signs and symptoms in breast |
| N830 | Follicular cyst of ovary |
| N831 | Corpus luteum cyst |
| N836 | Haematosalpinx |
| N837 | Haematoma of broad ligament |
| N838 | Other noninflammatory disorders of ovary, fallopian tube and broad ligament |
| N898 | Other specified noninflammatory disorders of vagina |
| N908 | Other specified noninflammatory disorders of vulva and perineum |
| N921 | Excessive and frequent menstruation with irregular cycle |
| N922 | Excessive menstruation at puberty |
| N923 | Ovulation bleeding |
| N924 | Excessive bleeding in the premenopausal period |
| N930 | Postcoital and contact bleeding |
| N938 | Other specified abnormal uterine and vaginal bleeding |
| N939 | Abnormal uterine and vaginal bleeding, unspecified |
| N950 | Postmenopausal bleeding |
| O208 | Other haemorrhage in early pregnancy |
| O209 | Haemorrhage in early pregnancy, unspecified |
| O441 | Placenta praevia with haemorrhage |
| O469 | Antepartum haemorrhage, unspecified |
| O679 | Intrapartum haemorrhage, unspecified |
| O695 | Labour and delivery complicated by vascular lesion of cord |
| O717 | Obstetric haematoma of pelvis |
| O720 | Third-stage haemorrhage |
| O721 | Other immediate postpartum haemorrhage |
| O722 | Delayed and secondary postpartum haemorrhage |
| O901 | Disruption of perineal obstetric wound |
| O902 | Haematoma of obstetric wound |
| P021 | Fetus and new-born affected by other forms of placental separation and haemorrhage |
| P100 | Subdural haemorrhage due to birth injury |
| P101 | Cerebral haemorrhage due to birth injury |
| P102 | Intraventricular haemorrhage due to birth injury |

| ICD-10 | ICD10Name |
|---|---|
| P103 | Subarachnoid haemorrhage due to birth injury |
| P109 | Unspecified intracranial laceration and haemorrhage due to birth injury |
| P120 | Cephalhaematoma due to birth injury |
| P269 | Unspecified pulmonary haemorrhage originating in the perinatal period |
| P510 | Massive umbilical haemorrhage of new-born |
| P519 | Umbilical haemorrhage of new-born, unspecified |
| P523 | Unspecified intraventricular (nontraumatic) haemorrhage of fetus and new-born |
| P524 | Intracerebral (nontraumatic) haemorrhage of fetus and new-born |
| P528 | Other intracranial (nontraumatic) haemorrhages of fetus and new-born |
| P529 | Intracranial (nontraumatic) haemorrhage of fetus and new-born, unspecified |
| P540 | Neonatal haematemesis |
| P542 | Neonatal rectal haemorrhage |
| P543 | Other neonatal gastrointestinal haemorrhage |
| P544 | Neonatal adrenal haemorrhage |
| P545 | Neonatal cutaneous haemorrhage |
| P546 | Neonatal vaginal haemorrhage |
| P549 | Neonatal haemorrhage, unspecified |
| P580 | Neonatal jaundice due to bruising |
| P581 | Neonatal jaundice due to bleeding |
| R040 | Epistaxis |
| R041 | Haemorrhage from throat |
| R042 | Haemoptysis |
| R048 | Haemorrhage from other sites in respiratory passages |
| R049 | Haemorrhage from respiratory passages, unspecified |
| R18 | Ascites |
| R195 | Other faecal abnormalities |
| R233 | Spontaneous ecchymoses |
| R31 | Unspecified haematuria |
| R571 | Hypovolaemic shock |
| R58 | Haemorrhage, not elsewhere classified |
| S000 | Superficial injury of scalp |
| S001 | Contusion of eyelid and periocular area |
| S002 | Other superficial injuries of eyelid and periocular area |
| S003 | Superficial injury of nose |
| S004 | Superficial injury of ear |
| S005 | Superficial injury of lip and oral cavity |
| S007 | Multiple superficial injuries of head |
| S008 | Superficial injury of other parts of head |
| S013 | Open wound of ear |
| S019 | Open wound of head, part unspecified |
| S050 | Injury of conjunctiva and corneal abrasion without mention of foreign body |
| S051 | Contusion of eyeball and orbital tissues |

| ICD-10 | ICD10Name |
|---|---|
| S063 | Focal brain injury |
| S064 | Epidural haemorrhage |
| S065 | Traumatic subdural haemorrhage |
| S066 | Traumatic subarachnoid haemorrhage |
| S068 | Other intracranial injuries |
| S098 | Other specified injuries of head |
| S100 | Contusion of throat |
| S101 | Other and unspecified superficial injuries of throat |
| S141 | Other and unspecified injuries of cervical spinal cord |
| S241 | Other and unspecified injuries of thoracic spinal cord |
| S271 | Traumatic haemothorax |
| S272 | Traumatic haemopneumothorax |
| S278 | Injury of other specified intrathoracic organs |
| S279 | Injury of unspecified intrathoracic organ |
| S301 | Contusion of abdominal wall |
| S302 | Contusion of external genital organs |
| S341 | Other injury of lumbar spinal cord |
| S361 | Injury of liver or gallbladder |
| S368 | Injury of other intra-abdominal organs |
| S369 | Injury of unspecified intra-abdominal organ |
| S370 | Injury of kidney |
| S378 | Injury of other pelvic organs |
| S390 | Injury of muscle and tendon of abdomen, lower back and pelvis |
| S400 | Contusion of shoulder and upper arm |
| S408 | Other superficial injuries of shoulder and upper arm |
| S500 | Contusion of elbow |
| S501 | Contusion of other and unspecified parts of forearm |
| S600 | Contusion of finger(s) without damage to nail |
| S601 | Contusion of finger(s) with damage to nail |
| S701 | Contusion of thigh |
| S800 | Contusion of knee |
| S801 | Contusion of other and unspecified parts of lower leg |
| S901 | Contusion of toe(s) without damage to nail |
| S902 | Contusion of toe(s) with damage to nail |
| T009 | Multiple superficial injuries, unspecified |
| T060 | Injuries of brain and cranial nerves with injuries of nerves and spinal cord at neck level |
| T090 | Superficial injury of trunk, level unspecified |
| T093 | Injury of spinal cord, level unspecified |
| T140 | Superficial injury of unspecified body region |
| T144 | Injury of nerve(s) of unspecified body region |
| T145 | Injury of blood vessel(s) of unspecified body region |
| T146 | Injury of muscles and tendons of unspecified body region |

| ICD-10 | ICD10Name |
|---|---|
| T794 | Traumatic shock |
| T810 | Haemorrhage and haematoma complicating a procedure, not elsewhere classified |
| T811 | Shock during or resulting from a procedure, not elsewhere classified |
| T876 | Other and unspecified complications of amputation stump |
| T905 | Sequelae of intracranial injury |
| | Subgaleal hemorrhage |
| | Intracranial hemorrhage |

# 10.3.6. Variables for subgroup analysis

| Subgroups | ICD10<br>code | Standard<br>disease code | Note |
|---|---|---|---|
| Hypertension | | | Refer to 10.3.1 |
| Liver dysfunction | | | Refer to 10.3.1 |
| Renal impairment | | | Refer to 10.3.1 |
| | A162 | | Include only tubercular hemoptysis |
| | A165 | | Include only tubercular hemothorax |
| | B303 | | |
| | D500 | | |
| | D62 | | |
| | D66 | | Include only hemophiliac bleeding |
| | D683 | | Include only hemorrhagic disorder due to circulating anticoagulants |
| | D698 | | |
| | D699 | | |
| | E078 | | Include only tyroid bleeding |
| | E274 | | Include only adrenal bleeding |
| | G361 | | |
| Bleeding history | G951 | | Include only hematomyelia, spinal subdural hemorrhage,<br>hematorrhachis, spinal epidural hemorrhage and spontaneous<br>Cervical Epidural Hematoma |
| | G968 | | Include only spinal subarachnoid hemorrhage |
| | H052 | | Include only orbital fat hemorrhage |
| | H113 | | |
| | H168 | | Include only Hemorrhagic keratitis |
| | H208 | | Include only hemorrhagic iritis |
| | H210 | | |
| | H313 | | |
| | H350 | | Include only hemorrhagic retinitis and juvenile recurrent vitreoretinal hemorrhage |
| | H356 | | |
| | H357 | | Include only hemorrhagic retinal pigment epithelial detachment |
| | H405 | | Include only hemorrhagic glaucoma |
| | H431 | | , 5 5 |

| Subgroups ICD10 code | Standard<br>disease code | Note |
|---|---|---|
| H448 | | Include only intraocular hemorrhage |
| H470 | | Include only optic disc hemorrhage and optic nerve sheath |
| | | hemorrhage |
| H603 | | Include only otitis externa hemorrhagica |
| H669 | | Include only hemorrhagic otitis media |
| H738 | | Include only eardrum bleeding |
| H922 | | |
| I213 | | Include only Atrial thrombus as current complication |
| <u> </u> | | following acute myocardial infarction |
| <u> 1230</u><br><u>1312</u> | | |
| 1600<br>I600 | | |
| I601 | | |
| 1602 | | |
| <u>1602</u> | | |
| <u> 1604</u> | | |
| 1605 | | |
| I606 | | |
| I607 | | |
| I608 | | |
| I609 | | |
| I610 | | |
| <u> I611</u> | | |
| <u>I613</u> | | |
| <u>I614</u> | | |
| <u>I615</u> | | |
| <u>I616</u> | | |
| <u>I618</u> | | |
| <u>I619</u> | | |
| <u>I620</u> | | |
| <u> 1621</u><br>1629 | | |
| 1629<br>1638 | | Inculde only hemorrhagic cerebral infarction |
| 1690 | | miculde only hemorrhagic cereoral inharction |
| I691 | | |
| 1780 | | |
| 1788 | | |
| I850 | | |
| I864 | | Include only gastric variceal bleeding |
| J041 | | Include only hemorrhagic tracheitis |
| J339 | | Include only bleeding polyp |
| J90 | | Include only hemorrhagic pleural effusion |
| J942 | | |
| J950 | | Include only bleeding from a tracheostomy site |
| K049 | | Include only hemorrhage in the pulp |
| K068 | | Include only gingival hemorrhage |
| K121 | | Include only hemorrhagic stomatitis |
| K137 | | Include only oral hemorrhage |

ICD10 Standard **Subgroups** Note code disease code K148 Include only tongue root submucosal bleeding K226 K228 Include only esophageal hemorrhage K250 K252 K254 K256 K260 Exclude acute gastroduodenal mucosal lesion K262 K264 K266 K284 K290 K571 Include only Duodenal diverticulum bleeding K573 Include only bleeding from Sigmoid diverticulum, Transverse colon diverticulum, Descending colon diverticulum, Ascending colon diverticulum and Large intestine diverticulum K625 Include only Hemorrhoidal external hemorrhoids, K649 Hemorrhoids and Hemorrhoidal internal hemorrhoids K661 K762 K768 Include only hepatorrhagia K859 Include only acute hemorrhagic necrotizing pancreatitis K920 K921 K922 L508 Include only hemorrhagic urticaria M2506 M2509 N029 N288 Include only perirenal bleeding, nephrorrhagia and idiopathic hematuria N300 Include only acute hemorrhagic cystitis N304 Include only radiation-induced hemorrhagic cystitis N309 Include only hemorrhagic cystitis N328 Include only bladder hemorrhage N368 Include only urethremorrhagia N421 N488 Include only penile hemorrhage Include only Scrotal hemorrhage and Spermatic cord N501 hematoma

#### PFIZER CONFIDENTIAL

cyst

N645 N830

N831

N836

Include only thelorrhagia

Exclude luteal cyst

Include only follicular hemorrhage and hemorrhagic follicular

| Subgroups ICD10 code | Standard<br>disease code | Note |
|---|---|---|
| N837 | | |
| N838 | | Include only ovarian hemorrhage |
| N898 | | Include only vaginal hematoma |
| N908 | | Include only vulval hemorrhage |
| N921 | | |
| N922 | | |
| N923 | | |
| N924 | | |
| N930 | | |
| N938 | | |
| N939 | | |
| N950 | | |
| O717 | | |
| O901 | | |
| O902 | | |
| R040 | | |
| R041 | | |
| R042 | | |
| _R048 | | |
| R049 | | |
| R18 | | Include only hemorrhagic ascites |
| R195 | | Include only fecal occult blood |
| R233 | | |
| R31 | | |
| R571 | | Include only hemorrhagic shock |
| R58 | | |
| S000 | | Include only ecchymoma, hematoma and hemorrhage |
| S001 | | Include only hematoma and hemorrhage |
| S002 | | Include only hematoma |
| S003 | | Include only hematoma and hemorrhage |
| S004 | | Include only hematoma and hemorrhage |
| S005 | | Include only hematoma and hemorrhage |
| S007 | | Include only hematoma and hemorrhage |
| S008 | | Include only hematoma |
| S013 | | Include only hemorrhage |
| S050 | | Include only Corneal hematoma |
| S051 | | Include only traumatic vitreous hemorrhage and traumatic |
| | | hyphema |
| S063 | | Include only hematoma and hemorrhage |
| S064 | | |
| S065 | | |
| S066 | | |
| S068 | | Include only hematoma, hemorrhage |
| S098 | | Include only hemorrhage |
| S100 | | Include only hematoma |
| S101 | | |
| S141 | | Include only hematoma |
| S241 | | Include only hematoma |

| Subgroups | ICD10 | Standard | Note |
|---|---|---|---|
| Subgroups | code | disease code | 11010 |
| | S271 | | |
| | S272 | | |
| | S278 | | Include only hematoma |
| | S279 | | Include only hematoma |
| | S301 | | Include only hematoma |
| | S302 | | Include only hematoma |
| | S341 | | Include only hematoma |
| | S361 | | Include only hematoma |
| | S368 | | Include only hemorrhage |
| | S369 | | Include only hematoma |
| | S370 | | Include only hematoma |
| | S378 | | Include only hemorrhage |
| | S390 | | Include only hematoma |
| | S400 | | Include only hematoma |
| | S408 | | Include only hematoma |
| | S500 | | Include only hematoma |
| | S501 | | Include only hematoma |
| | S600 | | Include only hematoma |
| | S601 | | Include only hematoma |
| | S701 | | Include only hematoma |
| | S800 | | Include only hematoma |
| | S801 | | Include only hematoma |
| | S902 | | Include only hematoma |
| | T009 | | Include only hematoma and hemorrage |
| | T060 | | Include only spinal subarachnoid hemorrhage |
| | T090 | | Including only hematoma |
| | T093 | | Including only hematoma |
| | T140 | | Including only hematoma |
| | T144 | | Include only traumatic hematomyelia |
| | T145 | | Include only traumatic arterial hematoma |
| | T146 | | Include only Intramuscular hematoma |
| | T794 | | Include only traumatic hemorrhagic shock |
| | T810 | | Include only hematoma and hemorrage |
| | T811 | | Include only hemorragic shock |
| | T876 | | Include only hematoma |
| | T905 | | Include only sequelae after |
| Hemorrhage stroke | | | Refer to 10.3.1 |
| | E244 | | |
| | E52 | | Include only Alcoholic pellagra |
| | F100 | | |
| | G312 | | |
| Alaahal ahusa | G405 | | Include only alcoholic epilepsy |
| Alcohol abuse | G621 | | |
| | G701 | | Include only alcoholic neuropathy |
| | G721 | | |
| | H470 | | Include only alcoholic optic neuropathy |
| | I426 | | |
| | 1420 | | |

| Subgroups | ICD10<br>code | Standard<br>disease code | Note |
|---|---|---|---|
| | K292 | | |
| | K70 | | |
| | K852 | | |
| | K860 | | |
| | T519 | | |
| Antiplatelet drug | | | Refer to 5.4 |
| NSAIDs | | | Refer to 5.4 |
| | F54 | | Include only psychogenic gastric ulcer |
| | K221 | | |
| | K227 | | Include only Barrett's esophagus |
| | K25 | | |
| Peptic ulcer | K26 | | |
| replie dicei | K27 | | |
| | K28 | | |
| | K51 | | |
| | K626 | | |
| | K633 | | |
| Active cancer | | | Refer to 10.3.1 |
| Diabetes mellitus | | | Refer to 10.3.1 |
| Polypharmacy | | | Refer to 5.4 |